CLINICAL TRIAL: NCT00778362
Title: Splenic Function After Spleen-Preserving Distal Pancreatectomy With Excision of Splenic Artery and Vein
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yu-Wen Tien/Association Proferssor , Department of Surgery, National Taiwan University Hospital
Other Study IDs: 200805057R
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Overwhelming Post-Splenectomy Infection
Keywords: OPSI; Splenectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Splenectomy: all patients received splenectomy (patient list will be applied from Dept. of Pathology) at National Taiwan University Hospital in the last 20 years.

SUMMARY:
The spleen may be removed due to benign hematologic disorders, such as idiopathic thrombocytopenic purpura and hereditary spherocytosis, or malignancies, such as lymphomas and leukemias. Splenectomy may also be performed due to splenic traumas or in association of some surgical procedures, when combined splenectomy will make the operations easier. The most well known procedure is distal pancreatectomy combined with splenectomy.

In this research, there are two main goals. Firstly, establish the data about the incidence of overwhelming postsplenectomy infection (OPSI) in our country. Currently, the western data of the incidence, morbidity rate and mortality rate of OPSI is well established and vaccination along with prophylactic antibiotics is strongly recommended. Since the incidence of OPSI in our country isn't clear, most (>95%) splenectomized patients in our hospital (National Taiwan University Hospital) did not have vaccination or prophylactic antibiotics. We'll try to determine the incidence of OPSI by reviewing of our hospital charts and by structured interviews with patients.

The spleen is a phagocytic filter. So asplenic patients have higher risks of getting infection and some spleen-preserving procedures are proposed. In our initial experiences, distal pancreatectomy with splenic artery and vein divided could be safely performed and greatly increased the possibility of preservation of spleen. However, when the spleen was preserved with dividing the splenic artery and vein, the blood supply to the spleen will be shifted from splenic artery to short gastric artery. Although a substantial immunologic advantage exists if splenic tissue remains, this may not offer sufficient protection from encapsulated bacteria if splenic arterial blood flow is reduced because experimental animal studies have demonstrated that an intact splenic arterial system is necessary for optimal control of infection. Thus, although the spleen is preserved in above mentioned procedure, the function of the preserved spleen is questionable and has never been studied of. Our second object is to determine the splenic function after after spleen-preserving distal pancreatectomy with excision of splenic artery and vein by comparison of abdominal computed tomography and immunological function of patients before and after operation. Besides, we'll designed an animal experiment to examine the rate of pneumococcal clearance by the spleen and to determine the relationship between splenic blood flow and splenic tissue mass in bacterial clearance from the blood when the splenic vessels were divided.

ELIGIBILITY:
Inclusion Criteria:

* all patients received splenectomy (patient list will be applied from Dept. of Pathology) at National Taiwan University Hospital in the last 20 years.

Exclusion Criteria:

* who rejected interview.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients received splenectomy (patient list will be applied from Dept. of Pathology) at National Taiwan University Hospital in the last 20 years.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
A questionnaire will be administered to assess 1. the degree of knowledge and patient compliance and their role in the prevention of OPSI; 2. history of vaccination and prophylactic antibiotics to prevent OPSI; 3. infection episodes after splenectomy. | twenty year after operation

SECONDARY OUTCOMES:
to determine the benefits (preserved immunologic function) and risk (gastric varices and even bleeding) of preservation of spleen after distal pancreatectomy without conservation of splenic artery | every one year after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Wen Tien, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan